

Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Investigate the Immunogenicity and Safety of Subcutaneous Administration of a Tetravalent Dengue Vaccine Candidate in Healthy Adolescent Subjects in Non-Endemic Area(s) for Dengue

SAP Approve Date: 30 January 2019

NCT Number: NCT03341637

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable (PPD) information or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



#### STATISTICAL ANALYSIS PLAN

STUDY NUMBER: DEN-315

A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Investigate the Immunogenicity and Safety of Subcutaneous Administration of a Tetravalent Dengue Vaccine Candidate in Healthy Adolescent Subjects in Non-Endemic Area(s) for Dengue

Immunogenicity and Safety of TDV in Adolescents in Non-Endemic Area(s)

#### PHASE 3

Version: Final, 1.0

Date: 30 January 2019

| Prepared by: |
|--------------|
| PPD |

Based on:

Protocol Version: 2.0

1D + 00 I

Protocol Date: 09 January 2018

#### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

# 1.1 Approval Signatures

Electronic signatures can be found on the last page of this document.

# 2.0 TABLE OF CONTENTS

| 1.0 TITLE PAGE | 1 |
|----------------------------------------------------------|------|
| 1.1 Approval Signatures | 2 |
| 2.0 TABLE OF CONTENTS | 3 |
| 3.0 LIST OF ABBREVIATIONS | 5 |
| 4.0 OBJECTIVES | 6 |
| 4.1 Primary Objective | 6 |
| 4.2 Secondary Objectives | 6 |
| 4.3 Additional Objectives | 6 |
| 4.4 Study Design | 6 |
| 5.0 ANALYSIS ENDPOINTS | 8 |
| 5.1 Primary Endpoint | 8 |
| 5.2 Secondary Endpoints | 8 |
| 6.0 DETERMINATION OF SAMPLE SIZE | 9 |
| 7.0 METHODS OF ANALYSIS AND PRESENTATION | 10 |
| 7.1 General Principles | 10 |
| 7.1.1 Data Presentation | 10 |
| 7.1.2 Study Day, Baseline and Analysis Window Definition | ıs10 |
| 7.1.3 Handling of Missing Data | 12 |
| 7.1.4 Implausible Values | 13 |
| 7.2 Analysis Sets | 13 |
| 7.3 Disposition of Subjects | 15 |
| 7.4 Demographic and Other Baseline Characteristics | 15 |
| 7.5 Medical History and Concurrent Medical Conditions | 15 |
| 7.6 Medication History and Concomitant Medications | 16 |
| 7.7 Investigational Product Exposure and Compliance | 16 |
| 7.8 Efficacy Analysis | 16 |
| 7.9 Pharmacokinetic/Pharmacodynamic Analysis | 16 |
| 7.10 Other Outcomes | 17 |
| 7.10.1 Primary Immunogenicity Analyses | 17 |
| 7.10.2 Secondary Immunogenicity Analyses | 17 |
| 7.11 Safety Analysis | 18 |
| 7.11.1 Adverse Events | 18 |
| 7.11.2 Clinical Laboratory Evaluations | 21 |
| 7.11.3 Vital Signs | 21 |

| 7.11.4 | 12-Lead ECGs | 21 |
|---|---|---|
| | Other Observations Related to Safety | |
| | terim Analysis | |
| | hanges in the Statistical Analysis Plan | |
| | RENCES | |
| LIST OF IN | -TEXT TABLES | |
| Table 7.a | Analysis Visit Windows | 11 |
| Table 7.b | Plausible Data Ranges | |
| Table 7.c | Criteria for Exclusion from the PPS | |
| Table 7.d | Overview of Unsolicited Adverse Events | 21 |
| Table 8.a | Schedule of Trial Procedures | 24 |
| Table 8.b | Solicited Local (Injection Site) and Systemic AEs | 26 |
| Table 8.c | Severity of Solicited Safety Parameters | |
| LIST OF IN | -TEXT FIGURES | |
| Figure 4.a | Schematic of Trial Design | 7 |
| LIST OF AF | PPENDICES | |
| Appendix A | Schedule of Trial Procedures | 24 |
| Appendix B | Solicited Local (Injection Site) and Systemic Adverse Events and Severity | 26 |

#### 3.0 LIST OF ABBREVIATIONS

AE Adverse event
BMI Body mass index
CRF Case Report Form
FAS Full analysis set
GMT Geometric mean titer

ICH International Conference on Harmoniyation

IP Investigational product

LAR Legally authorized representative

LLOD Lower limit of detection
LLOQ Lower limit of quantification

M0, 3, 4, 9 Month 0, 3, 4, 9

MAAE Medically attended adverse event

MedDRA Medical Dictionary for Regulatory Activities

MNT<sub>50</sub> Microneutralization test 50%

PPS Per-protocol set
PT Preferred term

SAE Serious adverse event
SAP Statistical analysis plan
SAS Statistical analysis system

SC Subcutaneous

SOC System organ class

TDV Tetravalent dengue vaccine candidate

WHO Drug World Health Organization Drug Dictionary

#### 4.0 OBJECTIVES

# 4.1 Primary Objective

• To describe the neutralizing antibody response against each dengue serotype at 1 month post second dose of a tetravalent dengue vaccine candidate (TDV) or placebo in dengue-naive adolescent subjects.

# 4.2 Secondary Objectives

## <u>Immunogenicity:</u>

- To describe the persistence of the immune response at 6 months post second dose of TDV or placebo in dengue-naive adolescent subjects.
- To describe the seropositivity rates for all dengue serotypes at 1 month and 6 months post second dose of TDV or placebo in dengue-naive adolescent subjects, where seropositivity is defined as a reciprocal neutralizing titer ≥10.

#### Safety:

• To describe the safety profile following a first and second dose of TDV or placebo at Day 1 (Month 0 [M0]) and Day 90 (Month 3 [M3]), respectively.

#### 4.3 Additional Objectives

Not applicable.

## 4.4 Study Design

This is a randomized, double-blind, placebo-controlled, phase 3 trial in 400 healthy adolescent subjects aged 12 to 17 years in a non-endemic country(ies) for dengue with 2 parallel groups to investigate the immunogenicity and safety of subcutaneous (SC) administration of a 2 dose regimen of TDV.

Subjects will be randomized in a 3:1 ratio (TDV [300 subjects]: placebo [100 subjects]) using an interactive response technology, as follows:

- Group 1: SC administration of TDV at Day 1 (M0) and Day 90 (M3).
- Group 2: SC administration of placebo at Day 1 (M0) and Day 90 (M3).

The trial duration for each subject will be approximately 270 days (9 months) including trial dose administration (Day 1 [M0] and Day 90 [M3]) and follow-up through Day 270 [Month 9 (M9)].

A schematic of the trial design is included in Figure 4.a. A schedule of trial procedures is provided in Appendix A.





M=Month, V=Visit

# <u>Immunogenicity evaluation:</u>

Dengue neutralizing antibodies (microneutralization test 50% [MNT<sub>50</sub>]) will be measured using blood samples collected from all subjects at pre-first dose (Day 1 [M0]), and at 1 month and 6 months post second dose (Day 120 [Month 4 (M4)]) and Day 270 [M9], respectively).

#### Safety evaluation:

- Diary cards will be distributed for the recording of:
  - Solicited local (injection site) adverse events (AE) for 7 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination+6 subsequent days). These will include: injection site pain, injection site erythema, and injection site swelling.
  - Solicited systemic AEs for 14 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination+13 subsequent days). These will include: fever, headache, asthenia, malaise, and myalgia.
- Unsolicited AEs for 28 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination+27 subsequent days).
- Serious adverse events (SAE) and medically attended adverse events (MAAE) for the trial duration. MAAEs are defined as AEs leading to a medical visit to or by a healthcare professional, including visits to an emergency department, but not fulfilling seriousness criteria.

Data collection will be by electronic Case Report Form (CRF).

#### 5.0 ANALYSIS ENDPOINTS

# 5.1 Primary Endpoint

• Geometric mean titers (GMT) of neutralizing antibodies (MNT<sub>50</sub>) for each of the 4 dengue serotypes at 1 month post second dose (Day 120 [M4]).

# 5.2 Secondary Endpoints

#### <u>Immunogenicity:</u>

- GMTs of neutralizing antibodies (MNT<sub>50</sub>) for each of the 4 dengue serotypes at 6 months post second dose (Day 270 [M9]).
- Seropositivity rates (% of subjects seropositive) for each of the 4 dengue serotypes at 1 month and 6 months post second dose (Day 120 [M4]) and Day 270 [M9], respectively).
- Seropositivity rates (% of subjects seropositive) for multiple (2, 3, or 4) dengue serotypes at 1 month and 6 months post second dose (Day 120 [M4]) and Day 270 [M9], respectively).

Note: Seropositivity is defined as a reciprocal neutralizing titer  $\geq 10$ .

#### Safety:

- Frequency and severity of solicited local (injection site) AEs for 7 days (day of vaccination+6 subsequent days) and solicited systemic AEs for 14 days (day of vaccination+13 subsequent days) after each TDV/placebo dose on Day 1 (M0) and Day 90 (M3).
- Percentage of subjects with any unsolicited AEs for 28 days (day of vaccination+27 subsequent days) after each TDV/placebo dose on Day 1 (M0) and Day 90 (M3).
- Percentage of subjects with MAAEs and SAEs and throughout the trial.

# 6.0 DETERMINATION OF SAMPLE SIZE

As the analysis of this trial is descriptive and is not based on testing formal null hypotheses, the sample size was not determined based on formal statistical power calculations. The sample size is considered sufficient to address the objectives of the trial.

#### 7.0 METHODS OF ANALYSIS AND PRESENTATION

# 7.1 General Principles

This statistical analysis plan (SAP) was developed based on the information provided in Protocol DEN-315, Version 2.0 dated 09 January 2018 [1] and on International Conference on Harmonization (ICH) E3 [2] and E9 [3] Guidelines.

All statistical analyses will be generated using the statistical analysis system SAS® Version 9.2 or higher.

The SAP provides details regarding the definition of analysis variables and analysis methodology to address all trial objectives. No inferential analyses will be performed for this trial, ie, all analyses described in this SAP will be exploratory only.

A blinded data review will be conducted prior to unblinding of subject's trial group assignment. This review will assess the accuracy and completeness of the trial database, subject evaluability, and appropriateness of the planned statistical methods.

#### 7.1.1 Data Presentation

In general, descriptive summaries will be provided by trial group.

Unless specified otherwise, number of subjects with non-missing observations, mean or geometric mean, SD or geometric SD, median, minimum, and maximum will be presented for continuous data. Frequency and percent will be presented for categorical data. In summary tables for categorical data for which categories are defined on the CRF, all categories will be presented as specified, even if the subject count within that category is zero. For other categorical data (eg, AEs and medications/vaccinations), only categories with at least one subject will be presented.

Minimum and maximum values will be presented using the same number of decimal places as the recorded data. Means, geometric means, and medians will be presented to 1 more decimal place than the recorded data. SD and geometric SD will be presented to 2 more decimal places than the recorded data, with possible exceptions made for derived data. The CI about a parameter estimate will be presented using the same number of decimal places as the parameter estimate (ie, 1 more decimal place than the recorded data). Percentages will be presented to 1 decimal place (eg, 80.3%).

All data collected will be presented in listings, sorted by trial group, site number, subject number, and date/time of the finding, if applicable. If not stated otherwise, screen failure subjects will be grouped and listed at the end.

#### 7.1.2 Study Day, Baseline and Analysis Window Definitions

Study Day 1 (M0) is defined as the date of the first trial vaccination, as recorded on the CRF vaccination form. Other study days are defined relative to Study Day 1 (M0), with Day -1 being the day prior to Day 1 (M0).

Baseline is defined as the last non-missing measurement taken before the first trial vaccination. Where time is available, the time of data collection must be prior to the first trial vaccination time. Day 1 (M0) observations taken after the first trial vaccination are considered post-Baseline values.

A windowing convention for immunogenicity and safety (vital signs) data will be used to determine the analysis value of a variable for a given trial visit. Following the schedule of trial procedures (Appendix A), analysis visit windows will be calculated relative to the days when each trial dose was administered (Day 1 [M0] and Day 90 [M3]).

If more than one measurement for a variable is obtained for a subject within the same visit window, the measurement with the date closest to the scheduled visit date will be used. In the event that 2 measurements within a given visit window are equidistant to the scheduled visit date, the later observation will be used. Both scheduled and unscheduled visits will be considered equally for the visit mapping for both immunogenicity and safety (vital signs) data.

The analysis visit windows for each trial visit are displayed in Table 7.a.

**Table 7.a** Analysis Visit Windows

| | | | Analysis Visit Windows | |
|---|---|---|---|---|
| Visit | Scheduled<br>Visit Day<br>(Month) | Scheduled<br>Vaccination | Full Analysis Set & Safety Set | Per-Protocol Set |
| V1 | Day 1 (M0) | Dose 1 | Prior [≤1 day] (a) to Dose 1 | Prior [≤1 day] (a) to Dose 1 |
| V2 | Day 30 | | 2 – 60 <sup>(b)</sup> days after Dose 1 | Not applicable (no blood sample |
| | (M1) | | (applies to Safety Set only) | is taken at V2) |
| V3 | Day 90<br>(M3) | Dose 2 | 61 – 115 <sup>(b)</sup> days after Dose 1 and Prior [≤1 day] <sup>(a)</sup> to Dose 2 | Not applicable (no blood sample is taken at V3) |
| | | | (applies to Safety Set only) | |
| V4 | Day 120<br>(M4) | | 2 – 105 <sup>(b)</sup> days after Dose 2 or<br><u>Safety Set:</u><br>116 – 195 <sup>(b)</sup> days after Dose 1 <sup>(c)</sup> | 29 – 37 <sup>(b)</sup> days after Dose 2 |
| | | | Full Analysis Set:<br>2 – 195 <sup>(b)</sup> days after Dose 1 <sup>(c)</sup> | |
| V5 | Day 270<br>(M9) | | ≥106 <sup>(b)</sup> days after Dose 2 or<br>≥196 <sup>(b)</sup> days after Dose 1 <sup>(c)</sup> | 173 – 194 <sup>(b)</sup> days after Dose 2 |

<sup>(</sup>a) Blood draw for immunogenicity assessments and assessment of vital signs must be prior to the vaccination scheduled for the same visit, and where time is available, the time of the blood/vital signs collection must be prior to the vaccination time. Day 1 (M0) observations taken after the first trial vaccination are considered post-Baseline values.

<sup>(</sup>b) Number of days after the visit is calculated with 1 day increment. For example, for V2 number of days after V1 is calculated as [Date of V2] – [Date of V1] + 1 (day).

<sup>(</sup>c) Applies to subjects who missed the second dose at V3.

#### 7.1.3 Handling of Missing Data

Data will be presented in the listings as reported. For the summaries and analysis, the following conventions apply.

# Immunogenicity data

Dengue neutralizing antibody titers (MNT $_{50}$ ) which are below the lower limit of detection (LLOD, 10) will be imputed with a value of 5 (half of the LLOD). If a reported value is between the LLOD and the lower limit of quantification (LLOQ, which differs between serotypes), this value will be imputed with the mid-point between the LLOD and LLOQ. For example, given a LLOQ of 18 for a serotype, all values between 10 and 18 will be imputed with 14 for this serotype.

No imputation methods will be used for missing immunogenicity data and all analyses will be based on complete records only.

#### Adverse event data

Missing information regarding 'relationship to investigational product (IP)' (related/not related) for solicited systemic and unsolicited AEs and 'severity' (mild/moderate/severe) for unsolicited AEs will be handled using the worst-case approach. Thus, unsolicited AEs with missing severity will be considered as 'severe' and solicited systemic and unsolicited AEs with missing relationship will be considered as 'related'.

Missing and partial unsolicited AE start dates may be imputed only to determine the temporal relationship between the start date of the event and the dose date of the most appropriate vaccination that the AE should be allocated with (ie, Vaccination 1 or Vaccination 2). An AE should be temporally allocated with the correct dose using the following rules:

- If the AE start and end dates are both completely missing, the AE will be allocated with the first trial vaccination;
- If at least month and/or the year of the AE start is/are available, the AE will be allocated with the latest vaccination prior to the AE start date;
- If the AE start date is completely missing, or the available start date information is insufficient to distinguish between the 2 trial vaccinations, but an AE end date or a partial AE end date (ie, month and/or year) is available, the AE end date will be assessed and the AE will be allocated with the vaccination after which the event ends. This is based on the assumption that any AE starting after Vaccination 1 and ongoing on the day of Vaccination 2 would be identified during the clinical assessments that are performed before administration of the second trial vaccination. If partial end date information indicates possible association with both vaccinations, the AE will be allocated with the first trial vaccination.

#### Prior/concomitant medication/vaccination data

Missing and partial medication/vaccination dates will be assessed only to distinguish between a prior or a concomitant medication/vaccine. A medication will be considered prior only if the partial end date indicates that it was stopped before first trial vaccination. A vaccine will be considered prior only if the partial vaccination date indicates that it was given before the first trial vaccination. In all other cases the medication or vaccine will be considered concomitant.

# Medical history/concurrent medical conditions

In case the "End Date" or "End Date Unknown" fields are missing on the medical history/concurrent medical conditions form of the CRF and from the partial date it can't be concluded that the event is clearly a medical history, the event will be considered concurrent medical condition

# 7.1.4 Implausible Values

Data outside the plausible ranges as defined in will be excluded from respective analyses, but presented as recorded in data listings including a flag that highlights implausible values.

| | Parameter | Applicable age range | Plausible range |
|---|---|---|---|
| Demographic/ | Height | 12 – 17 years | 100 – 210 cm |
| Physical examination | Weight | 12 – 17 years | 20 - 200 kg |
| Solicited AEs | Erythema | ≥ 6 years | ≤ 500 mm |
| | Swelling | ≥ 6 years | ≤ 500 mm |
| | Body Temperature (a) | All ages | 32-43°C |
| Vital Signs | Heart Rate | All ages | 40 – 200 beats/min |
| | Systolic Blood Pressure | All ages | 70-180 mmHg |
| | Diastolic Blood Pressure | All ages | 30-120 mmHg |
| | Respiratory Rate | All ages | 5 – 80 breaths/min |

<sup>(</sup>a) Also applicable to body temperature measurements collected as vital signs.

#### 7.2 Analysis Sets

**Randomized Set**: The Randomized Set will consist of all randomized subjects, regardless of whether any dose of IP (TDV or placebo) was received.

Subjects will be summarized according to the IP they are randomized to.

**Safety Set**: The Safety Set will consist of all randomized subjects who received at least 1 dose of IP.

Subjects will be summarized according to the IP they received. For example, a subject randomized to TDV but vaccinated with placebo will be analyzed in the TDV group. Subjects who received different IPs at first and second vaccinations (eg, subject vaccinated with TDV at

first vaccination and with placebo at second vaccination) will be considered in a separate group. Data for this group, labelled as "Unplanned IP sequence", will be displayed in selected summaries and all listings (including subject mappings for AEs) generated for the Safety Set.

**Full Analysis Set (FAS)**: The FAS will consist of all randomized subjects who received at least 1 dose of the IP and for whom a valid a pre-dose (Baseline) measurement and at least 1 valid post-dose measurement is available for immunogenicity.

Subjects will be summarized according to IP they are randomized to.

**Per-Protocol Set (PPS)**: The PPS will exclude all subjects seropositive to any serotype of dengue virus at Baseline (Seropositivity is defined as a reciprocal neutralizing titer  $\geq 10$ .) and will include all subjects in the FAS who have no major protocol violations.

The criteria (ie, the major protocol violations) as described in Table 7.c will be used to identify subjects who will be excluded from the PPS and will be identified prior to database lock and unblinding of subject's trial group assignment. These criteria are considered to have a potentially significant impact on the immunogenicity results of the subject. Subjects excluded from the PPS due to receiving an incorrect IP will be identified after unblinding.

Table 7.c Criteria for Exclusion from the PPS

| Criteria for Exclusion | Probable Method of Identification |
|---|---|
| Not receiving at least one dose of the IP (a) | Identified programmatically using dosing data |
| Not having a valid pre-dose (Baseline) and at least 1 valid post-dose measurement <sup>(b)</sup> | Identified programmatically using immunogenicity data |
| Subjects seropositive to any serotype of dengue neutralizing titers at Baseline (Day 1 [M0]) | Identified programmatically using immunogenicity data |
| Not receiving both doses of the IP | Identified programmatically using dosing data |
| Receiving the second trial vaccination inadmissibly outside of the scheduled visit window (ie, outside Day 90 [-15/+25 days]) | Identified programmatically using dosing data |
| Receiving the incorrect IP(s) for vaccination 1 and/or vaccination 2 | Identified after unblinding |
| Product preparation error | Identified through protocol deviation log |
| Subject meets any of the following exclusion criteria: 6, 7, 9, 10, 11, 12, 15, 19, 20, 21 | Identified programmatically using CRF-recorded data; Identified through protocol deviation review/medical review |
| Use of prohibited medications/vaccines | Identified through medical review based on CRF-recorded data |

<sup>(</sup>a) Subjects with this protocol violation will be excluded from the Safety Set, and thus also from the FAS and the PPS.

<sup>(</sup>b) Subjects with this protocol violation will be excluded from the FAS, and thus also from the PPS.

# 7.3 Disposition of Subjects

Trial information will be presented for all screened subjects, including the date the first subject signed the informed consent form, the date of the first subject's first visit, the date of the last subject's last visit, the date of first subject's first vaccination, the date of last subject's first vaccination, the date of last subject's second vaccination, the Medical Dictionary for Regulatory Activities (MedDRA) version, the World Health Organization Drug Dictionary (WHODrug) version, and the SAS version used for analysis.

Disposition of all screened subjects will be summarized descriptively, including a summary of the number of screened subjects, the number of randomized subjects and the primary reason for not being eligible for randomization. The number of screen failures and their characteristics will also be summarized.

Disposition for all randomized subjects will be summarized by trial group. Disposition categories include:

- Number of subjects randomized by trial site.
- Number of subjects randomized, but not vaccinated (including primary reason for being randomized, but not vaccinated).
- Number of subjects in the Randomized Set, Safety Set, FAS, and PPS.
- Number of subjects who completed the vaccine regimen/trial visits.
- Number of subjects who prematurely discontinued the vaccine regimen/trial visits.
- Primary reason for premature discontinuation of the vaccine regimen/trial visits.

Additionally, significant protocol deviations as captured on the CRF will be summarized based on the Safety Set.

#### 7.4 Demographic and Other Baseline Characteristics

Age, gender, race, and other Baseline characteristics will be summarized descriptively based on the Safety Set, FAS and PPS.

#### 7.5 Medical History and Concurrent Medical Conditions

Medical history and concurrent medical conditions will be coded according to the MedDRA coding system. The version of the dictionary used will be specified in the CSR.

A medical history is defined as any significant condition/disease that stopped at or prior to first dose of IP. A concurrent medical condition is defined as any significant condition/disease that is ongoing at the time the first dose of IP is administered.

Summary tables will be provided by SOC and PT based on the Safety Set.

## 7.6 Medication History and Concomitant Medications

Medication history, vaccine history, concomitant medications, and concomitant vaccines will be coded according to WHODrug. The version of the dictionary used will be specified in the CSR.

A prior medication/vaccine (history) is any medication/vaccine which intake was stopped before first dose of IP. A concomitant medication/vaccine is any medication/vaccine ongoing at the time the first dose of IP is administered, or taken/administered on/after the first dose of IP.

Summary tables for medication history and concomitant medications will be provided by Anatomical Therapeutic Chemical class level 2 and preferred medication name. Vaccine history and concomitant vaccines will be summarized by vaccine type and name as recorded on the CRF. Summaries will be provided based on the Safety Set.

# 7.7 Investigational Product Exposure and Compliance

The Investigator records all injections of the IP given to the subject on the CRF.

Investigational product compliance will be summarized by trial group (including a separate group of subjects who received different IPs at first and second vaccination [if any]) for the Safety Set presenting the number and percentage of subjects receiving:

- 1) First vaccination only
- 2) Both vaccinations

The duration of follow-up after the first dose of IP (defined as the number of days from first vaccination to end of the trial) will be summarized by trial group for the Safety Set as a continuous variable (number of subjects [n], mean, SD, median, minimum, and maximum), and also as categorical variable (frequency and percentage of subjects) for the following intervals: 1-30 days, 31-90 days, 91-120 days, 121-270 days, 121-270 days. Additionally, the duration of follow-up after the second dose of IP (defined as the number of days from second vaccination to end of the trial) will be summarized in a similar way as a continuous variable and also as categorical variable for the following intervals: 1-30 days, 1-90 days, 1-180 days, 1-180 days.

#### 7.8 Efficacy Analysis

Not applicable.

# 7.9 Pharmacokinetic/Pharmacodynamic Analysis

Not applicable.

#### 7.10 Other Outcomes

# 7.10.1 Primary Immunogenicity Analyses

The primary immunogenicity endpoint of this trial is the GMTs of dengue neutralizing antibodies (derived from dengue MNT<sub>50</sub> results) for each of the 4 dengue serotypes 1 month post second dose (ie, Day 120 [M4]).

The number of subjects with non-missing assessments, geometric mean with 95% CI, geometric SD, median, minimum and maximum will be presented for neutralizing antibody titers for each dengue serotype by trial group. GMTs will be calculated as anti-logarithm of  $\Sigma$ (log transformed titer/n), where n is the number of subjects with titer information. The 95% CI for GMTs will be calculated as the anti-log transformation of upper and lower limits for a 2-sided CI of the mean of the log-transformed titers (based on student's t-distribution).

The primary immunogenicity endpoint will be summarized by trial group based on the PPS. A supportive analysis will be provided using the FAS.

#### 7.10.2 Secondary Immunogenicity Analyses

The secondary immunogenicity endpoints of this trial are:

- GMTs of neutralizing antibodies (MNT<sub>50</sub>) for each of the 4 dengue serotypes at 6 months post second dose (ie, Day 270 [M9]).
- Seropositivity rates (% of subjects seropositive) for each of the 4 dengue serotypes at 1 month and 6 months post second dose (ie, Day 120 [M4]) and Day 270 [M9], respectively).
- Seropositivity rates (% of subjects seropositive) for multiple (2, 3, or 4) dengue serotypes at 1 month and 6 months post second dose (ie, Day 120 [M4]) and Day 270 [M9], respectively).

GMTs of dengue neutralizing antibodies (derived from dengue MNT<sub>50</sub> results) at 6 months post second dose will be analyzed in analogy to the primary immunogenicity endpoint.

For the seropositivity rates for each dengue serotype, the percentage of subjects seropositive along with exact 2-sided 95% CI will be presented by trial group and visit. The exact 2-sided 95% CI of seropositivity rate will be calculated based on Clopper-Pearson method [4]. Seropositivity is defined as a reciprocal neutralizing titer ≥10.

Seropositivity rates for multiple dengue serotypes will be analyzed in analogy to the seropositivity rates for each dengue serotype, as described above, and will include the percentage of subjects with:

- monovalent seropositivity (seropositive for only 1 of the 4 dengue serotypes),
- bivalent seropositivity (seropositive for any 2 of the 4 dengue serotypes),
- trivalent seropositivity (seropositive for any 3 of the 4 dengue serotypes),
- tetravalent seropositivity (seropositive for all 4 dengue serotypes),

- at least bivalent seropositivity (seropositive for  $\geq 2$  dengue serotypes),
- at least trivalent seropositivity (seropositive for  $\geq 3$  dengue serotypes)

The secondary immunogenicity endpoints will be summarized by trial group based on the PPS. Supportive analyses will be provided based on the FAS.

In addition, GMTs (including 95% CIs) over time (all visits) and reverse cumulative distribution curves (all visits except baseline) will be plotted (line plots) by dengue serotype, trial group and visit based on the PPS. Seropositivity rates will be graphically presented by dengue serotype, for at least trivalent, and for tetravalent seropositivity, and by trial group and visit using bar graphs including the percentage of subjects seropositive and corresponding 95% CIs.

#### 7.11 Safety Analysis

All summaries of safety data will be based on subjects in the Safety Set.

#### 7.11.1 Adverse Events

Unless otherwise specified, AEs will be summarized by trial group after first trial vaccination, second trial vaccination, and any trial vaccination.

## Reactogenicity (Solicited AEs)

Solicited AEs are collected for at least 30 min after each vaccination at the site (in-clinic assessment). In addition, subjects are provided with a diary card for the recording of solicited local (injection site) AEs, including injection site pain, injection site erythema, and injection site swelling, for 7 days following vaccination (day of vaccination + 6 days). Subjects are also provided with a diary card for the recording of solicited systemic AEs (fever, headache, asthenia, malaise, and myalgia) for 14 days following vaccination (day of vaccination + 13 days). For the local (injection site) AEs erythema and swelling, the subject/the subject's legally authorized representative (LAR) will record the length of the longest diameter in mm. However, for the analysis these data will be displayed in cm. For the systemic AE fever, the subject/the subject's LAR will record the body temperature in either °F or °C. For the analysis, all data will be displayed in °C. Severity grades for erythema and swelling will be derived from the recorded diameters, and fever will be presented using the proposed temperature increments published by the Brighton Collaboration Fever Working Group [5]. Details of solicited local (injection site) and systemic AEs, and severity of solicited safety parameters are given in Appendix B.

Missing data for solicited AEs will not be imputed unless otherwise specified in Section 7.1.3. For each trial group and solicited AE, the denominator for the percentage will exclude subjects with completely missing data (ie, subject does not have at least 1 recorded result [ie, none, mild, moderate, or severe]) for the solicited AE in the period being summarized.

For each solicited AE, the number and the percentage of subjects reporting an event will be summarized by event severity for the following intervals post-vaccination:

- 30 minutes (in-clinic assessment of solicited local [injection site] and systemic AEs analyzed separately from diary-recorded solicited AEs)
- Within 7 days (solicited local [injection site] AEs)
- Within 14 days (solicited systemic AEs)
- Days 1 7 (daily, solicited local [injection site] AEs)
- Days 1 14 (daily, solicited systemic AEs)
- Days 1 3 and Days 4 7 (solicited local [injection site] AEs)
- Days 1 7 and Days 8 14 (solicited systemic AEs)

For subjects with more than 1 episode of the same event, the maximum severity will be used for tabulations.

For solicited systemic AEs, the number and percentage of subjects will also be summarized by relationship to IP (assessed by the Investigator) for the following intervals post-vaccination:

- 30 minutes
- Within 14 days

Subjects will only be counted once if the subject has more than 1 episode of the same event. In the case where the subject has both related and unrelated solicited systemic AEs, the subject will be counted under the related category. All solicited local (injection site) AEs are considered as related to IP.

A summary of the day of first onset of each event and the number of days subjects reported each event will be presented post-vaccination. The number of days a subject reported each event is calculated as the total of all days the subject reported the event, regardless of whether the event was reported on consecutive days.

An overview table for solicited AEs post-vaccination will be provided including:

- 30 minutes in-clinic assessment (solicited local [injection site] and systemic AEs combined)
- Solicited AEs (solicited local [injection site] and systemic AEs combined)
- Solicited local [injection site] AEs
- Solicited systemic AEs (overall and by relationship to IP)
- Prolonged solicited AEs (overall and for solicited local [injection site] and systemic AEs separately)

Prolonged solicited AEs that continue beyond Day 7 (for local [injection site] AEs) or Day 14 (for systemic AEs) will be captured on the AE CRF with appropriate indication ("continued solicited AE"). These prolonged solicited AEs will be presented in separate listings and will not be included in any unsolicited AE summary or listing.

#### **Unsolicited AEs**

Unsolicited AEs will be assessed for 28 days following administration of each trial dose (day of vaccination + 27 subsequent days). MAAEs, SAEs and AEs leading to IP withdrawal or trial discontinuation will be collected from first trial dose (Day 1 [M0]) until the end of the trial (Day 270 [M9]). Unsolicited AEs, MAAEs, SAEs, and AEs leading to IP withdrawal or trial discontinuation will be coded according to the current version of MedDRA and summarized by SOC and PT.

In general, the number of events, number of subjects, and the percentage of subjects will be tabulated by trial group at each of the following levels: overall summary (any AEs/subjects with any AEs) and by SOC and PT. Subjects reporting more than 1 occurrence for the term (level) being summarized will be counted only once in the number/percentage of subjects. Percentages will be based on the number of subjects in the Safety Set who received the respective trial dose.

Unsolicited AEs up to 28 days post-vaccination will be summarized as follows:

- By SOC and PT;
- By SOC and PT including events with frequency greater than 2% in any trial group;
- By SOC and PT including non-serious events with frequency greater than 2% in any trial group (including a separate group of subjects who received different IPs at first and second vaccination [if any]);
- By SOC and PT for IP related events;
- By SOC and PT for IP related events with frequency greater than 2% in any trial group;
- By SOC, PT, and severity (mild, moderate, severe).

MAAEs post-vaccination throughout the trial duration will be summarized as follows:

- By SOC and PT;
- By SOC and PT for IP related events;
- By SOC, PT, and severity (mild, moderate, severe).

SAEs post-vaccination throughout the trial duration will be summarized as follows:

- By SOC and PT (including a separate group of subjects who received different IPs at first and second vaccination [if any]);
- By SOC and PT for IP related events.

AEs leading to IP withdrawal or trial discontinuation post-vaccination throughout the trial duration will be summarized as follows:

• By SOC and PT (including a separate group of subjects who received different IPs at first and second vaccination [if any]);

#### • By SOC and PT for IP related events.

In addition, overview tables by trial group will be generated for unsolicited AEs (collected up to 28 days post-vaccination), SAEs, MAAEs and AEs leading to IP withdrawal or trial discontinuation including the variables as outlined in Table 7.d.

**Table 7.d Overview of Unsolicited Adverse Events** 

| | All AEs<br>(28 days post-<br>vaccination) | SAEs | MAAEs | AEs leading to<br>IP withdrawal<br>and/or trial<br>discontinuation |
|---|---|---|---|---|
| Relationship to IP | ✓ | ✓ | ✓ | ✓ |
| Relationship to trial procedure | ✓ | ✓ | ✓ | ✓ |
| Severity | ✓ | ✓ | ✓ | ✓ |
| AEs leading to IP withdrawal and/or trial discontinuation | ✓ | ✓ | ✓ | |
| AEs leading to IP withdrawal | ✓ | ✓ | ✓ | ✓ |
| AEs leading to trial discontinuation | ✓ | ✓ | ✓ | ✓ |
| MAAEs | ✓ | | | ✓ |
| SAEs and<br>Non-serious AEs | <b>√</b> | | | ✓ |
| Deaths | ✓ | ✓ | | ✓ |

Subject mappings (ie, list of subject numbers in each category of SOC and PT, and each trial group) will be provided for unsolicited AEs, SAEs, MAAEs and AEs leading to IP withdrawal or trial discontinuation.

#### 7.11.2 Clinical Laboratory Evaluations

Not applicable.

#### 7.11.3 Vital Signs

The vital signs collected in the trial include systolic and diastolic blood pressure, heart rate, body temperature, height, weight, and body mass index (BMI). Summary statistics (number of subjects [n], mean, SD, median, minimum, and maximum) will be presented by trial group and visit (observed data and changes from Baseline).

#### 7.11.4 12-Lead ECGs

Not applicable.

#### 7.11.5 Other Observations Related to Safety

Not applicable.

# 7.12 Interim Analysis

No interim analysis is planned for this trial.

# 7.13 Changes in the Statistical Analysis Plan

The SAP contains no changes to the planned analyses described in the protocol.

#### 8.0 REFERENCES

- 1. A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Investigate the Immunogenicity and Safety of Subcutaneous Administration of a Tetravalent Dengue Vaccine Candidate in Healthy Adolescent Subjects in a Non-Endemic Area(s) for Dengue. Takeda Vaccines, Inc. Protocol No. DEN-315, Version 2.0, dated 09 January 2018.
- 2. ICH Harmonized Tripartite Guideline Clinical Trial Reports: Structure and Content, E3 (http://www.ich.org/products/guidelines/efficacy/efficacy-single/article/structure-and-content-of-clinical-study-reports.html).
- 3. ICH Harmonized Tripartite Guideline Statistical Principles for Clinical Trials, E9 (http://www.ich.org/products/guidelines/efficacy/efficacy-single/article/statistical-principles-for-clinical-trials.html).
- 4. Clopper CJ and Pearson ES. The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrika. 1934;26: 404-13.
- 5. Marcy SM, Kohl KS, Dagan R, Nalin D, Blum M, Jones MC, et al. Fever as an adverse event following immunization: case definition and guidelines of data collection, analysis and presentation. Vaccine. 2004;22(5-6):551-6.

# **Appendix A** Schedule of Trial Procedures

**Table 8.a** Schedule of Trial Procedures

| Visit number | V1 | V2 | V3 | V4 | V5 (a) |
|---|---|---|---|---|---|
| | Day 1 | Day 30 | <b>Day 90</b> | Day 120<br>(V3+30 days) | Day 270<br>(V3+180 days) |
| Day | M0 | <b>M1</b> | <b>M3</b> | M4 | M9 (ET) |
| Visit window (days) | ±0 | -1/+7 | -4/+7 | -1/+7 | -7/+14 |
| Informed consent/assent (b) | X | | | | |
| Assessment of eligibility criteria (c) | X | | | | |
| Demographics | X | | | | |
| Medical history | X | | | | |
| Concomitant medications/vaccinations (d) | X | X | X | X | X |
| Check criteria for delay of trial vaccination | X | | X | | |
| Check contraindications to trial vaccination | | | X | | |
| Complete physical examination (e) | | | X | | |
| Targeted physical examination (f) | | X | | X | X |
| Vital signs (g) | X | X | X | X | X |
| Pregnancy test (h) | X | | X | | |
| Pregnancy avoidance guidance (i) | X | X | X | X | |
| Randomization | X | | | | |
| Blood sample for dengue neutralizing antibodies (5 mL) <sup>(j)</sup> | X | | | X | X |
| Trial dose administration (k) | X | | X | | |
| Injection site evaluation (1) | X | | X | | |
| Distribution | X | | X | | |
| Diary card (m) Review/collection | | X | | X | |
| Unsolicited adverse events (AE) (n) | X | X | X | X | |
| Serious adverse events (SAE) and AEs leading to subject discontinuation or withdrawal (o) | X | X | X | X | X |
| Medically attended AEs (MAAE) (o) | X | X | X | X | X |

ET=Early Termination; M=month; V=visit

<sup>(</sup>a) If the subject terminates early, Day 270 (M9) procedures should be performed.

<sup>(</sup>b) Up to 28 days prior to the day of randomization.

<sup>(</sup>c) Review of inclusion/exclusion criteria will be performed prior to administration of the first trial dose at Day 1 (M0). After eligibility is assessed and written informed consent/assent has been obtained, subjects will be randomized to receive either 2 doses of TDV or placebo by subcutaneous (SC) injection.

<sup>(</sup>d) Any other vaccination against any flavivirus (licensed or investigational, including any other dengue vaccine) during the entire trial period, all concomitant medications, vaccine history from 1 month (minimum 28 days) prior to administration of each trial dose of TDV or placebo up to 1 month (minimum 28 days) thereafter, steroids and immunostimulants within 60 days prior to Day 1 (M0), immunoglobulins and blood products within 3 months prior to Day 1 (M0), and immunosuppressive therapy within 6 months prior to Day 1 (M0).

- (e) Physical examination including measurement of vital signs (see footnote [g]), weight and height; body mass index (BMI) will be calculated automatically. Measurement of height is only required at Day 1 (M0).
- (f) Subjects may undergo a brief symptom-directed physical examination. Clinically significant changes from the Baseline examination should be recorded in the subject's source documents and electronic Case Report Form (CRF).
- (g) Vital signs including (but not limited to) the measurement of systolic blood pressure, diastolic blood pressure, heart rate, and body temperature.
- (h) Pregnancy testing (serum or urine) for females of childbearing potential. Results must be confirmed and documented as negative prior to each trial dose administration. Additional pregnancy tests may be performed during the trial if deemed necessary by the Investigator. Females of childbearing potential who are sexually active will be reminded during trial visits to adhere to acceptable contraceptive methods up to 6 weeks after the last dose of IP (Day 90 [M3]).
- (i) Females of childbearing potential who are sexually active will be provided with information on acceptable methods of contraception as part of the subject informed consent/assent process and will be asked to sign a consent form/assent form stating that they understand the requirements for avoidance of pregnancy and donation of ova. Subjects will be reminded during trial visits to adhere to acceptable contraceptive methods and not to donate ova up to 6 weeks after the last dose of IP (Day 90 [M3]).
- (j) The blood sample at Day 1 (M0) should be taken prior to administration of the first trial dose. The blood sample at Visit 4 (Day 120 [M4]) should be taken at least 28 days after the second trial dose at Day 90 (M3).
- (k) TDV (Group 1) or placebo (Group 2).
- (1) Injection site assessed by trial staff for pain, erythema, and swelling for at least 30 minutes following administration of each trial dose.
- (m) Diary cards will be distributed for the collection of 1) solicited local (injection site) AEs for 7 days following administration of each trial dose (including the day of administration), and 2) solicited systemic AEs for 14 days following administration of each trial dose (including the day of administration).

  The Investigator will categorize all events by severity (mild, moderate or severe), and will assess causality to trial dose administration for solicited systemic events (related or not related).
- (n) Unsolicited AEs will be collected for 28 days following administration of each trial dose (including the day of administration) by interview. The Investigator will categorize events by severity (mild, moderate or severe) and will assess causality to trial dose administration (related or not related).
- (o) MAAEs, SAEs, and AEs leading to subject discontinuation or withdrawal will be collected for the trial duration. The Investigator will categorize all events by severity (mild, moderate or severe) and will assess causality to trial dose administration (related or not related).

# Appendix B Solicited Local (Injection Site) and Systemic Adverse Events and Severity

Table 8.b Solicited Local (Injection Site) and Systemic AEs

| Solicited local (injection site) AEs: | Pain |
|---------------------------------------|-----------|
| | Erythema |
| | Swelling |
| Solicited systemic AEs: | Fever (a) |
| | Headache |
| | Asthenia |
| | Malaise |
| | Myalgia |

<sup>(</sup>a) Fever is defined as a body temperature  $\ge 38^{\circ}$ C (100.4°F) regardless of the method used [5].

**Table 8.c** Severity of Solicited Safety Parameters

| Adverse Event | Severity grade | Severity |
|---|---|---|
| Pain at injection site | 0 | None |
| | 1 | Mild: No interference with daily activity |
| | 2 | Moderate: Interference with daily activity with or without treatment |
| | 3 | Severe: Prevents daily activity with or without treatment |
| Erythema at injection site (a) | 0 | < 25 mm |
| | 1 | Mild: $25 - \le 50 \text{ mm}$ |
| | 2 | Moderate: $> 50 - \le 100 \text{ mm}$ |
| | 3 | Severe: > 100 mm |
| Swelling at injection site (a) | 0 | < 25 mm |
| | 1 | Mild: $25 - \le 50 \text{ mm}$ |
| | 2 | Moderate: $> 50 - \le 100 \text{ mm}$ |
| | 3 | Severe: > 100 mm |
| Headache | 0 | None |
| | 1 | Mild: No interference with daily activity |
| | 2 | Moderate: Interference with daily activity with or without treatment |
| | 3 | Severe: Prevents normal daily activity with or without treatment |
| Asthenia | 0 | None |
| | 1 | Mild: No interference with daily activity |
| | 2 | Moderate: Interference with daily activity |
| | 3 | Severe: Prevents normal daily activity |
| Malaise | 0 | None |
| | 1 | Mild: No interference with daily activity |
| | 2 | Moderate: Interference with daily activity |
| | 3 | Severe: Prevents normal daily activity |
| Myalgia | 0 | None |
| | 1 | Mild: No interference with daily activity |
| | 2 | Moderate: Interference with daily activity |
| | 3 | Severe: Prevents normal daily activity |
| Fever (b) | NA | None |
| | NA | 38.0-<38.5°C |
| | NA | 38.5-<39.0°C |
| | NA | 39.0-<39.5°C |
| | NA | 39.5-<40.0°C |
| | NA | 40.0-<40.5°C |
| | NA | 40.5-<41.0°C |
| | NA | ≥41.0°C |

NA = not applicable

<sup>(</sup>a) Subjects are to record greatest surface diameter in mm on the diary card.

<sup>(</sup>b) Fever is defined as a body temperature  $\geq 38^{\circ}$ C (100.4°F) regardless of the method used [5].

# Signature Page for DEN-315 Statistical Analysis Plan Title:

| | PPD |
|----------|-----|
| Approval | |
| Approval | |
| Approval | |

Document Number: TAK-003-02463 v1.0